## Effects of Blood Orange Juice Consumption on Endothelial Function in Healthy Overweight/Obese Men and Premenopausal Women of European Origin

Date: January 10, 2017

Sixteen overweight/obese participants of European origin will be asked to consume blood orange juice and a control drink for 2 weeks in a random sequence, separated by a 1-week washout period. All measurements will be conducted prior to and following 2-week consumption. Subjects will be instructed to stay fasted and restrain from exercise for 12 hours before measurements in the morning. Anthropometric measures will be conducted. After the subject is supine and comfortable for 15 minutes to reach a cardiovascular steady state, blood pressure will be measured in triplicate with 2-minute intervals. Endothelial function will be evaluated via brachial artery FMD. Each test for a given subject will be performed at the same time of the day. Following brachial FMD measurement, venous blood samples from antecubital vein will be collected into vacutainers to produce serum and plasma. Spot urine samples will also be collected.